CLINICAL TRIAL: NCT04478071
Title: Vadadustat for the Prevention and Treatment of Acute Respiratory Distress Syndrome (ARDS) in Hospitalized Patients With Coronavirus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Akebia Therapeutics Inc. (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bentley J. Bobrow, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-20-0395; W81XWH-21-10032 (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Acute Respiratory Distress Syndrome; Coronavirus Infection
Keywords: COVID-19; ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome; Coronavirus Infections; COVID-19 | interventions — vadadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vadadustat (Experimental)
  Interventions: Drug: vadadustat
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vadadustat — Participants will receive vadadustat once daily for 14 days.
  Other Names: AKB-6548
  Arms: vadadustat
Drug: placebo — Participants will receive matching placebo once daily for 14 days.
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of vadadustat for the prevention and treatment of acute respiratory distress syndrome (ARDS) in hospitalized patients with Coronavirus Disease 2019 (COVID-19).

ELIGIBILITY:
Inclusion Criteria:

* Laboratory-confirmed diagnosis of COVID-19 by detection of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) RNA by Reverse transcription polymerase chain reaction (RT-PCR) from any specimen respiratory
* Admitted to the hospital within 36 hours
* Oxygen saturation of hemoglobin by pulse oximetry at room air ≤94%
* For patients admitted WITH respiratory symptoms, enrollment must occur within 36 hours of hospital admission. If the patient is admitted to the hospital with normal saturations, but develops respiratory symptoms DURING their hospital stay, enrollment may occur within 24 hours of desaturation to 94% or less on room air
* Understands the procedures and requirements of the study and provides written informed consent and authorization for protected health information disclosure

Exclusion Criteria:

* Hypersensitivity to vadadustat or any of its excipients
* Placed on mechanical ventilation before randomization
* Hemoglobin above the gender-specific upper limit of normal (ULN) at randomization: 16 g/dL for females and 18 g/dL for males
* Patients who have erythrocytosis or polycythemia vera
* Patient taking Probenecid, lopinavir or ritonavir
* Women who are pregnant or breastfeeding, or positive pregnancy test before randomization
* Patients not on maintenance dialysis with eGFC < 31 ml/min
* Patients who have received a solid organ transplant, heart, kidney, liver or lung
* Patients who are prisoners
* Patients who are currently Do Not Resuscitate (DNR) or Do Not Intubate (DNI)
* Patients with modified Rankin scale of 3 or greater
* Patient who are currently enrolled in any other interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2020-08-22 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bentley J. Bobrow, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vadadustat | Placebo
Started | 221 | 227
Completed Day 7 | 217 | 223
Completed Day 14 | 216 | 223
Completed Day 28 | 215 | 221
Completed | 215 | 221
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat | Placebo | Total
Number analyzed (Participants) | 221 | 227 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (14.8) | 50.7 (14.7) | 50.9 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 83 | 162
  Male | 142 | 144 | 286
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 158 | 151 | 309
  Not Hispanic or Latino | 63 | 76 | 139
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 26 | 47
  White | 168 | 170 | 338
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  United States | 221 | 227 | 448
Number of Participants with history of type 2 diabetes [Count of Participants; unit: Participants] | 62 | 73 | 135
Number of Participants with a history of hypertension [Count of Participants; unit: Participants] | 74 | 91 | 165
Body Mass Index [Median (Inter-Quartile Range); unit: kilograms per meter squared] — Population: Data were not collected for 3 participants in the placebo arm. Data were not collected for 3 participants in the vadadustat arm.
  kilograms per meter squared
    number analyzed (Participants) | 218 | 224 | 442
    (all) | 31.6 [27.0 to 36.2] | 32.8 [28.0 to 38.4] | 32.2 [27.5 to 37.9]
Days since onset of COVID symptoms [Median (Inter-Quartile Range); unit: days] — Population: Data were not collected for 8 participants in the placebo arm. Data were not collected for 5 participants in the vadadustat arm.
  days
    number analyzed (Participants) | 216 | 219 | 435
    (all) | 7 [5 to 10] | 7 [5 to 10] | 7 [5 to 10]
Score on the Modified Sequential Organ Failure Assessment (MSOFA) Scale [Mean (Standard Deviation); unit: score on a scale] — Modified Sequential Organ Failure Assessment (MSOFA) scale:
  Each of 5 organ systems is given a score of 0 to 4.The MSOFA scale total score is the sum of the score for the 5 organ systems. Total score ranges from 0 to 20, a higher score indicates a worse outcome. Discharged patients will be assigned a score of 0 and dead patients a score of 20.
  score on a scale | 2.73 (1.17) | 2.74 (1.19) | 2.73 (1.18)
Score on the National Institute of Allergy and Infectious Disease Ordinal Scale (NIAID-OS) [Mean (Standard Deviation); unit: score on a scale] — NIAID-OS:
  8 - Death 7 - Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation 6 - Hospitalized, on non-invasive ventilation or high flow oxygen devices 5 - Hospitalized, requiring supplemental oxygen 4 - Hospitalized, not requiring supplemental oxygen - requiring ongoing care (COVID-19 related or otherwise) 3 - Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care 2 - Not hospitalized, limit on activities and/or requiring home oxygen 1 - Not hospitalized, no limits on activities
  score on a scale | 5.3 (0.5) | 5.3 (0.5) | 5.3 (0.5)
Oxygen Saturation to Fraction of Inspired Oxygen (SpO2/FiO2) Ratio [Mean (Standard Deviation); unit: SpO2/FiO2 Ratio] — SpO2 (oxygen saturation) is the percentage of oxygen in the blood. The fraction of inspired oxygen (FiO2) is the percentage of oxygen a person inhales.
  SpO2/FiO2 Ratio | 217.4 (91.8) | 224.1 (94.2) | 220.8 (93)
Score ≥ 4 on the Modified Sequential Organ Failure Assessment (MSOFA) Scale [1] [Count of Participants; unit: Participants] — Modified Sequential Organ Failure Assessment (MSOFA) scale:
  Each of 5 organ systems is given a score of 0 to 4.The MSOFA scale total score is the sum of the score for the 5 organ systems. Total score ranges from 0 to 20, a higher score indicates a worse outcome. Discharged patients will be assigned a score of 0 and dead patients a score of 20.
  Participants | 69 | 73 | 142

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Classified 8 (Dead), 7 (Hospitalized, on Invasive Mechanical Ventilation or ECMO), or 6 (Hospitalized, on Non-invasive Ventilation or High Flow Oxygen Devices) on the NIAID Ordinal Scale
Description: National Institute of Allergy and Infectious Disease Ordinal Scale (NIAID-OS):
  8 - Death 7 - Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) 6 - Hospitalized, on non-invasive ventilation or high flow oxygen devices 5 - Hospitalized, requiring supplemental oxygen 4 - Hospitalized, not requiring supplemental oxygen - requiring ongoing care (COVID-19 related or otherwise) 3 - Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care 2 - Not hospitalized, limitation on activities and/or requiring home oxygen
  1 - Not hospitalized, no limitations on activities
Time Frame: day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 216 | 223
Participants | 43 | 53
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Trial used Bayesian analysis for superiority. Hypothesis Testing for Primary Outcome: Among adult hospital admissions with lab-confirmed diagnosis of COVID-19, vadadustat 900 mg will demonstrate superiority to placebo as defined by a lower probability, at treatment day 14, of death (8) or hospitalization, on invasive mechanical ventilation or ECMO (7) or hospitalization, on non-invasive ventilation or high flow oxygen devices (6) on the NIAID-OS. See Statistical Analysis Plan for more details; Test type: Superiority; Risk Difference (RD) = -0.036, 95% CI 2-sided [-0.084 to 0.009] — Risk difference of Vadadustat relative to Placebo. Values under "confidence interval" reflect Bayesian 95% credible interval rather than frequentist confidence interval
Statistical Analysis 2: Comparison: Vadadustat vs Placebo; Test type: Superiority; Posterior Probability = 0.94 — Posterior probability of the risk difference of Vadadustat relative to Placebo

2. Secondary Outcome: Number of Participants With a Total Score of 0 on the Modified Sequential Organ Failure Assessment (MSOFA) Scale
Description: Modified Sequential Organ Failure Assessment (MSOFA) scale:
  Each of 5 organ systems is given a score of 0 to 4.The MSOFA scale total score is the sum of the score for the 5 organ systems. Total score ranges from 0 to 20, a higher score indicates a worse outcome. Discharged patients will be assigned a score of 0 and dead patients a score of 20.
Time Frame: day 14
Population: Data were not collected for 2 participants in the vadadustat arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Placebo
Number analyzed (Participants) | 214 | 223
Participants | 156 | 157
Statistical Analysis 1: Comparison: Vadadustat vs Placebo; Trial used Bayesian analysis for superiority. Hypothesis Testing for Secondary Outcome: Among adult hospital admissions with lab-confirmed diagnosis of COVID-19, vadadustat 900 mg will demonstrate superiority to placebo as defined by a higher probability, at treatment day 14, of recovery on the MSOFA scale (MSOFA = 0); Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.92 to 1.1] — Risk ratio of Vadadustat relative to Placebo. Values under "confidence interval" reflect Bayesian 95% credible interval rather than frequentist confidence interval
Statistical Analysis 2: Comparison: Vadadustat vs Placebo; Test type: Superiority; Posterior probability = 0.57 — Posterior probability of the risk ratio of Vadadustat relative to Placebo

3. Other Pre Specified Outcome: Score on the Modified Sequential Organ Failure Assessment (MSOFA) Scale
Description: Modified Sequential Organ Failure Assessment (MSOFA) scale:
  Each of 5 organ systems is given a score of 0 to 4, as detailed below. The MSOFA scale total score is the sum of the score for the 5 organ systems. Discharged patients will be assigned a score of 0 and dead patients a score of 20.
  * Respiratory oxygen saturation(SpO2)/concentration of oxygen that a person inhales(FiO2): 0 (> 400); 1 (≤ 400); 2 (≤ 315); 3 (≤ 235); 4 (≤ 150)
  * Liver: 0 (No scleral icterus or jaundice); 3 (Scleral icterus or jaundice)
  * Cardiovascular, hypotension: 0 (No hypotension); 1 (MAP < 70 mm Hg); 2 (Dopamine ≤ 5 or dobutamine any dose); 3 (Dopamine > 5, Epinephrine ≤ 0.1, Norepinephrine ≤ 0.1); 4 (Dopamine > 15, Epinephrine > 0.1, Norepinephrine > 0.1)
  * Central Nervous System (CNS), Glasgow Coma Score: 0 (15), 1 (13 - 14); 2 (10 - 12); 3 (6 - 9); 4 (< 6)
  * Renal, Creatinine mg/dL: 0 (< 1.2); 1 (1.2 - 1.9); 2 (2.0 - 3.4); 3 (3.5 - 4.9); 4 (> 5.0)
Time Frame: day 7
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Score on the Modified Sequential Organ Failure Assessment (MSOFA) Scale
Description: as for outcome 3
Time Frame: day 14
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Ventilator-free Survival
Time Frame: day 7
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Ventilator-free Survival
Time Frame: day 14
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Overall Survival
Time Frame: day 7
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Overall Survival
Time Frame: day 14
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Number of Participants With Hypotension
Description: Hypotension is defined as Mean Arterial Pressure (MAP) <70 mm Hg or requirement for inotropes or vasopressors to maintain blood pressure.
Time Frame: day 7
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Number of Participants With Hypotension
Description: as for outcome 9
Time Frame: day 14
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Participants With Acute Kidney Injury
Time Frame: day 7
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Participants With Acute Kidney Injury
Time Frame: day 14
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Time to Hospital Discharge
Time Frame: From the time of hospital admission to hospital discharge (about 7 days)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 28 days
Arm/Group | Vadadustat | Placebo
All-Cause Mortality (participants affected / at risk) | 19/221 | 19/227
Serious Adverse Events (participants affected / at risk) | 61/221 | 73/227
Other Adverse Events (participants affected / at risk) | 109/221 | 116/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vadadustat (N=221) | Placebo (N=227)
Acute kidney injury (Investigations) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4)
Alanine aminotransferase and aspartate aminotransferase increased (Hepatobiliary disorders) | 0 (0) | 2 (2)
Alanine aminotransferase and aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 4 (4) | 10 (10)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation with rapid ventricular response (Cardiac disorders) | 0 (0) | 4 (4)
Bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Fungemia (Infections and infestations) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemoglobin increased (Investigations) | 3 (3) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intermittent sinus pauses (Cardiac disorders) | 0 (0) | 1 (1)
Non-ST elevation myocardial infarction type 2 (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 24 (24) | 24 (25)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 6 (6) | 3 (3)
Worsening pneumonia (Infections and infestations) | 42 (42) | 59 (59)
Worsening pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Arterial thromboembolism (Vascular disorders) | 1 (1) | 0 (0)
Ascending cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation and atrial flutter with rapid ventricular response (Cardiac disorders) | 1 (1) | 0 (0)
Bilateral pneumothoraces (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine increased (Renal and urinary disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Ejection fraction decreased due to dilated cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Neck abscess (Infections and infestations) | 1 (1) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Severse sepsis with shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcus aureus bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vadadustat (N=221) | Placebo (N=227)
Alanine aminotransferase increased (Investigations) | 69 (70) | 51 (51)
Anemia (Blood and lymphatic system disorders) | 30 (30) | 38 (39)
Aspartate aminotransferase increased (Investigations) | 30 (30) | 32 (33)
Hyperkalemia (Metabolism and nutrition disorders) | 24 (27) | 21 (21)
Hypermagnesemia (Metabolism and nutrition disorders) | 17 (17) | 33 (34)
Hyperphosphatemia (Metabolism and nutrition disorders) | 4 (4) | 16 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 19 (20) | 19 (20)
Hypokalemia (Metabolism and nutrition disorders) | 19 (19) | 17 (17)
Hyponatremia (Metabolism and nutrition disorders) | 24 (26) | 34 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04478071/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04478071/ICF_001.pdf